CLINICAL TRIAL: NCT00858247
Title: Significance of Vitamin D Status in Obese Adolescents- A Pilot Study to Examine the Effect of Vitamin D3 Supplementation on Insulin Resistance and Cardiovascular Risk Factors
Brief Title: Effect of Vitamin D3 Supplementation on Insulin Resistance and Cardiovascular Risk Factors in Obese Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Thrasher Research Fund (Other)
Responsible Party: Seema Kumar, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-008743; UL1RR024150 (NIH)
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: vitamin D; Obesity; Insulin sensitivity; Adolescent Obesity
MeSH Terms: conditions — Obesity; Insulin Resistance; Pediatric Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3-low dose (Experimental): Vitamin D3 400 IU capsule, one capsule daily for 12 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3-high dose (Experimental): Vitamin D3 2000 IU capsule, one capsule daily for 12 weeks.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — One arm would receive vitamin D3 at a dose of 400 IU by mouth once daily for 12 weeks and the other arm would receive vitamin D3 as a single oral daily dose of 2000 IU for 12 weeks.

SUMMARY:
The prevalence of obesity has reached epidemic proportions nationally as well as internationally. Currently, 16 % of American adolescents are obese. In adults, obesity is a risk factor for vitamin D insufficiency and up to 80% of obese adults have been noted to vitamin D insufficient. In adults, low vitamin D status appears to be associated with the development of type 2 diabetes and metabolic syndrome. There is little information on the prevalence of vitamin D insufficiency and its implications in obese adolescents. Additionally, it is unknown whether treatment of vitamin D insufficiency in adolescents might result in improvement in insulin resistance, lipids and cardiovascular risk markers.

We hypothesize that vitamin D insufficiency correlates positively with insulin resistance and cardiovascular risk in obese adolescents and that vitamin D3 supplementation improves insulin resistance and cardiovascular risk factors in this population. The purpose of the study is to determine the impact of vitamin D3 supplementation on various parameters of insulin secretion, insulin action, lipids and C-reactive protein in obese adolescents.

DETAILED DESCRIPTION:
The problem of childhood obesity has reached epidemic proportions both nationally and internationally. The prevalence of obesity has tripled in the last three decades and currently 16 % of American adolescents are obese. Nearly 30% of obese adolescents demonstrate a metabolic syndrome characterized by insulin resistance and dyslipidemia. These abnormalities lead to the development of type 2 diabetes mellitus and to increased cardiovascular morbidity and mortality. Obesity is a well-known risk factor for vitamin D insufficiency and up to 80% of obese adults have been found to be insufficient in vitamin D. Observational studies in adults have shown consistent associations between low vitamin D status and prevalence of type 2 diabetes mellitus and metabolic syndrome. There is paucity of data on the prevalence of vitamin D insufficiency and its implications in obese adolescents. It is also not known whether treatment of vitamin D insufficiency in children or adults might result in improvement in insulin resistance and cardiovascular risk factors.

Hypotheses: We hypothesize that vitamin D insufficiency correlates positively with insulin resistance and cardiovascular risk in obese adolescents and that vitamin D3 supplementation decreases insulin resistance and cardiovascular risk factors in this population.

Objectives:

1. Determine if there is any correlation between serum 25(OH)D levels and homeostasis model assessment of insulin resistance (HOMA-IR), HDL cholesterol and C-reactive protein, in obese adolescents.
2. Study the impact of vitamin D3 supplementation on various parameters reflecting insulin action, secretion, lipids and C-reactive protein in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 12-18 years
2. BMI is at or greater than the 95th percentile for age and gender

Exclusion Criteria:

1. Subjects with 25 (OH)- D levels >100 ng/mL
2. Serum calcium >10.8 mg/dL
3. Current cancer
4. Those taking a multivitamin supplementation
5. Hepatic or renal disorders
6. Type 1 or type 2 diabetes mellitus.
7. Those receiving insulin, metformin or oral hypoglycemic medications

   * Use of glucocorticoids and anti-seizure medications in the previous 6 months
   * Malabsorption syndromes such as celiac disease

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Kumar, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Javed A, Vella A, Balagopal PB, Fischer PR, Weaver AL, Piccinini F, Dalla Man C, Cobelli C, Giesler PD, Laugen JM, Kumar S. Cholecalciferol supplementation does not influence beta-cell function and insulin action in obese adolescents: a prospective double-blind randomized trial. J Nutr. 2015 Feb;145(2):284-90. doi: 10.3945/jn.114.202010. Epub 2014 Dec 17. PMID 25644349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the Mayo Clinic in Rochester, Minnesota.
Groups:
- Vitamin D3-low Dose: Vitamin D3 400 IU capsule, one capsule daily
  Vitamin D3: One arm would receive vitamin D3 at a dose of 400 IU by mouth once daily for 12 weeks and the other arm would receive vitamin D3 as a single oral daily dose of 2000 IU for 12 weeks.
- Vitamin D3-high Dose: Vitamin D3 2000 IU capsule, one capsule daily
  Vitamin D3: One arm would receive vitamin D3 at a dose of 400 IU by mouth once daily for 12 weeks and the other arm would receive vitamin D3 as a single oral daily dose of 2000 IU for 12 weeks.
Period: Baseline Assessment
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Started | 25 | 26
Completed | 23 | 24
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Poor IV access | 1 | 0
Not completed — Protocol Violation | 0 | 1
Period: Week 12 Follow-up
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Started | 23 | 24
Completed | 23 | 23
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 47 Subjects started the study, but one subject in the Vitamin D3-high dose arm only completed one visit. The baseline characteristics are reported on the 47 subjects who started the study.
Groups:
- Vitamin D3-low Dose: Vitamin D3 400 IU capsule, one capsule daily
- Vitamin D3-high Dose: Vitamin D3 2000 IU capsule, one capsule daily
- Total: Total of all reporting groups
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.5 [13.5 to 16.6] | 14.7 [13.5 to 16.0] | 14.5 [13.5 to 16.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 18 | 27
  Male | 14 | 6 | 20
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Resistance After 12 Weeks of Vitamin D3 Supplementation
Description: Insulin resistance (IR) is a physiological condition in which cells fail to respond to the normal actions of the hormone insulin. The body produces insulin, but the cells in the body become resistant to insulin and are unable to use it as effectively, leading to hyperglycemia. Beta cells in the pancreas subsequently increase their production of insulin, further contributing to hyperinsulinemia.
  From the fasting glucose and insulin measurements, insulin resistance was calculated by the homeostasis model assessment of insulin resistance (HOMA -IR) as: HOMA -IR = fasting insulin concentration (µU/mL) x fasting glucose concentration (mmol/L)/22.5. High HOMA-IR scores denote increased insulin resistance.
Time Frame: Baseline, 12 weeks
Population: All subjects had blood drawn but some tests such as insulin could not be done in some cases due to sample issues. This lab test was calculated from other parameters and not drawn per se. If the values obtained did not allow a calculation of the lab test, then the results could not be reported.
Measure: Mean (Standard Deviation); unit: HOMA score
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Number analyzed (Participants) | 21 | 21
HOMA score | 0.01 (1.34) | -0.27 (4.95)
Statistical Analysis 1: Comparison: Vitamin D3-low Dose vs Vitamin D3-high Dose; Test type: Superiority or Other; p = 0.95, ANCOVA

2. Secondary Outcome: Change in Total Cholesterol After 12 Weeks of Vitamin D Supplementation
Description: Less than 200 mg/dL is desirable, >200 mg/dL is borderline high, >240 mg/dL is High
Time Frame: baseline, 12 weeks
Population: One subject in the high-dose arm dropped out before the week 12 assessment, so the reporting population on the high dose arm was 23, not 24.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Number analyzed (Participants) | 23 | 23
mg/dL | 4.7 (24.3) | 3.5 (16.8)
Statistical Analysis 1: Comparison: Vitamin D3-low Dose vs Vitamin D3-high Dose; Test type: Superiority or Other; p = 0.80, ANCOVA

3. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol After 12 Weeks of Vitamin D Supplementation
Description: LDL cholesterol is considered to be the main source of cholesterol buildup and blockage in the arteries. Less than 100 mg/dL is optimal, >130 mg/dL is borderline high, >160 mg/dL is high, >190 mg/dL is very high.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Number analyzed (Participants) | 23 | 23
mg/dL | 4.6 (22.0) | 1.3 (15.6)
Statistical Analysis 1: Comparison: Vitamin D3-low Dose vs Vitamin D3-high Dose; Test type: Superiority or Other; p = 0.65, ANCOVA

4. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol After 12 Weeks of Vitamin D Supplementation
Description: HDL (good) cholesterol protects against heart disease, so for HDL, higher numbers are better. A level less than 40 mg/dL is low and is considered a major risk factor because it increases your risk for developing heart disease. HDL levels of 60 mg/dL or more help to lower your risk for heart disease.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Number analyzed (Participants) | 23 | 23
mg/dL | 1.3 (6.8) | 1.9 (5.7)
Statistical Analysis 1: Comparison: Vitamin D3-low Dose vs Vitamin D3-high Dose; Test type: Superiority or Other; p = 0.68, ANCOVA

5. Secondary Outcome: Change in Triglycerides After 12 Weeks of Vitamin D Supplementation
Description: The current recommendation on fasting blood triglyceride levels: < 150 mg/dL is normal, >150 mg/dL is borderline high, and >200 mg/dL is high.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Number analyzed (Participants) | 23 | 23
mg/dL | -4.7 (56.7) | 1.7 (43.5)
Statistical Analysis 1: Comparison: Vitamin D3-low Dose vs Vitamin D3-high Dose; Test type: Superiority or Other; p = 0.40, ANCOVA

6. Secondary Outcome: Change in High-Sensitivity C-Reactive Protein After 12 Weeks of Vitamin D Supplementation
Description: The high-sensitivity C-reactive protein test measures your risk for heart problems. <1.0 mg/L is lowest risk, 1.0-3.0 mg/L is average risk, and >3.0 mg/L is highest risk.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Number analyzed (Participants) | 23 | 23
mg/L | -0.2 (1.2) | -0.5 (1.7)
Statistical Analysis 1: Comparison: Vitamin D3-low Dose vs Vitamin D3-high Dose; Test type: Superiority or Other; p = 0.47, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the duration of the study, an average of 12 weeks.
Arm/Group | Vitamin D3-low Dose | Vitamin D3-high Dose
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 1/23 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3-low Dose (N=23) | Vitamin D3-high Dose (N=24)
Lightheaded and dizzy (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No